CLINICAL TRIAL: NCT06831240
Title: New Rear Anti-tip Device for Manual Wheelchairs: Subjective Input from Wheelchair Service Providers and End-Users
Brief Title: New Rear Anti-tip Device for Manual Wheelchairs: Subjective Input (RAD-SI)
Acronym: RAD-SI
Status: Not yet recruiting | Type: Observational
Sponsor: Nova Scotia Health Authority (Other)
Responsible Party: Sponsor
Other Study IDs: WRT2025-RAD-SI
Record Dates: First submitted 2025-01-31; First posted 2025-02-18 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Wheelchair Users; Caregivers; Wheelchair Service Providers; Amputation; Stroke; Spinal Cord Injury
Keywords: wheelchair; rear anti-tip device
MeSH Terms: conditions — Stroke; Spinal Cord Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (3):
- Local wheelchair service providers: Wheelchair service providers will be Occupational Therapists or Occupational Therapy Assistants for the focus groups.
  Interventions: Other: Local wheelchair service provider questionnaires
- Global wheelchair service providers: For the online survey, participants will be people who self-identify as wheelchair service providers.
  Interventions: Other: Global wheelchair service provider questionnaires
- End-users: For end-users, we will study wheelchair users, in some cases with their caregivers.
  Interventions: Other: End-users questionnaires

INTERVENTIONS:
Other: Local wheelchair service provider questionnaires — The local wheelchair service providers will complete a questionnaire that includes demographic data, to allow us to describe the sample, and a questionnaire about rear anti-tip devices for manual wheelchairs.
  Groups: Local wheelchair service providers
Other: Global wheelchair service provider questionnaires — The global wheelchair service providers will complete a questionnaire that includes demographic data, to allow us to describe the sample, and a questionnaire about rear anti-tip devices for manual wheelchairs.
  Groups: Global wheelchair service providers
Other: End-users questionnaires — The end-users will complete a questionnaire that includes demographic and clnical data, to allow us to describe the sample, and a questionnaire about rear anti-tip devices for manual wheelchairs.
  Groups: End-users

SUMMARY:
The objective of this study is to obtain subjective input from wheelchair service providers and end-users about their experiences with conventional rear anti-tip devices (C-RADs) of manual wheelchairs and the potential usefulness of a new design.

DETAILED DESCRIPTION:
The limited safety and maneuverability afforded by conventional rear anti-tip devices (C-RADs) for manual wheelchairs and the inability of most wheelchair users to perform conventional wheelies both provided the incentive for designing a self-deploying rear anti-tip device (RAD) that appears to enhance both safety and performance. The principal feature of the device was an adjustable-arc arm. The outer end of the device was out of the way during normal wheelchair use but self-deployed when needed, making it suitable for long-term use. The axis of rotation of the anti-tip arm was above the rear-wheel axle. In the resting position, the arm angled downward and backward but did not need to extend past the rearmost dimension of the rear wheel. When the wheelchair tipped backward sufficiently, the lower end of the arm (on which a small swivel caster was located) contacted the ground. The force of the tipping chair rotated the arm through an arc (hence the name Arc-RAD) until it hit a cam that acted as a stop to prevent any further tipping of the wheelchair. When the wheelchair was upright, the wheelchair user could grasp a lever and switch among four cam settings without getting out of the chair, should a different arc occasionally be needed (e.g., to allow the increased arc needed to descend a steep incline). In the deployed position, the occupied wheelchair was extremely stable.

Proof-of-Concept Studies and Refinements. It was demonstrated that the Arc-RAD could provide both stability and wheelie-like function in seven studies. Although the Arc-RAD prototype that was used was suitable to confirm proof-of-concept, the investigators wished to overcome the design barriers that had been identified. Through iterative refinements, the investigators have overcome the major design barriers.

STATEMENT OF RESEARCH QUESTION

The objective of this study is to obtain subjective input from wheelchair service providers and end-users about their experiences with C-RADs of manual wheelchairs and the potential usefulness of the Arc-RAD.

RESEARCH PLAN

Study design. This is a non-interventional cross-sectional survey following the Strengthening the Reporting of Observational Studies in Epidemiology (STROBE) Guidelines. The investigators will use focus groups, an online survey to seek subjective input from wheelchair service providers and semi-structured interviews to seek subjective input from end-users.

Setting. The study will be based in Halifax at the Nova Scotia Rehabilitation and Arthritis Centre (NSRAC) Site.

Ethical Issues. Before proceeding, the study will have been approved by the Research Ethics Board of the Nova Scotia Health Authority. All participants will provide informed consent. For end-users who require caregiver assistance, caregivers will also complete an Informed Consent Form. For respondents to the online survey, participants will attest to an informed-consent statement to access the survey.

Participants. Wheelchair service providers will be Occupational Therapists or Occupational Therapy Assistants for the focus groups. For the online survey, participants will be people who self-identify as wheelchair service providers. For end-users, the investigators will study wheelchair users, stratified by a Wheelchair Skills Level Questionnaire (Version 5.4.2) into 3 groups of approximately equal size:

1. Wheelchair users who are caregiver-dependent for community skills (and their caregivers). Although a wheelchair user may have different people who serve from time to time in the caregiver capacity, for the purposes of this study the focus is on a single caregiver who has been identified by the wheelchair user and who meets the inclusion/exclusion criteria.
2. Wheelchair users who are independent for community skills but who are not wheelie-capable.
3. Wheelchair users who are independent for wheelie-dependent skills.

Sample Size. For the focus groups of wheelchair service providers, the investigators will continue to enroll participants until apparent saturation, expected to require no more than 20 wheelchair service providers. For the online data collection from wheelchair service providers, to provide sufficient data to be meaningful, the investigators will seek to obtain data from at least 100 wheelchair service providers globally. For the end-users, the investigators will study 30 wheelchair users and 10 caregivers. Sample sizes of 20 or fewer have commonly been used in similar studies.

Recruitment. The investigators expect to be able to recruit all focus-group and end-user participants from the Nova Scotia Rehabilitation and Arthritis Centre (NSRAC). Study advertisements will be used to complement recruitment. If the rate of participant accrual is insufficient, the investigators will extend the recruitment efforts to potential participants in other hospital sites, in the community and/or nursing-home settings. Potential wheelchair-service-provider participants for the focus groups will be approached by the Research Coordinator (a co-worker). Potential end-user participants will be approached by clinicians with whom the potential participants are working. Potential participants willing to learn more about the study will be informed about it by the Research Coordinator and screened by interview for inclusion/exclusion criteria. For potential wheelchair-using participants in Group 1 who meet the eligibility requirements, the Research Coordinator will contact and screen (remotely if necessary) the appropriate caregiver identified by the wheelchair-user. For CONSORT-reporting purposes, the investigators will describe potential participants who are screened, those recruited and drop-outs. Clinicians will be notified that the clients have been enrolled in the study.

For the online survey, the investigators will target self-identifying English-speaking wheelchair service providers around the world. The investigators will seek respondents to the survey through the Facebook page of the Wheelchair Skills Program, through snowball recruitment, as well as through the email distribution lists of organizations with international reach that are willing to assist.

Inclusion/Exclusion Criteria. All participants will be at least 18 years of age, willing to participate, alert, co-operative, able to see and hear the video demonstrations, able to communicate in English, have the capacity to provide informed consent and committed to setting a scheduled time for the study activity. Wheelchair service providers will be Occupational Therapists or Occupational Therapy Assistants who self-identify as being regularly involved in the wheelchair provision process. End users will be wheelchair users and, for those in Group 1, caregivers. Each wheelchair-using participant will be a person who has used a manual wheelchair for at least one month. Each caregiving participant will be a caregiver who spends an average total of at least 2 hours per week with the manual wheelchair user that includes manual wheelchair mobility. Caregiver or wheelchair-using participants will be excluded if there are emotional problems that might make participation unsafe or unpleasant. For the online survey, the investigators will include anyone who self-identifies as being regularly involved in the wheelchair provision process.

Questionnaires. There are three separate, but similar questionnaires. In each, demographic, clinical and/or wheelchair data will be collected to describe the participants. Subsequently for each group, a series of photographs and video recordings regarding rear anti-tip devices will be used to demonstrate the issue under consideration and pose the questions. For the video recordings of the Arc-RAD, the investigators used a rigid-frame manual wheelchair. For each of the potential uses of the Arc-RAD, the two questions shown in Table 1 will be asked.

Table 1. Questions regarding each potential use of the Arc-RAD

1. Comments or questions (if any)?
2. How useful does the participant think this feature would be?" (pick one score) Pick one Score Meaning 5 Extremely useful 4 Somewhat useful 3 Maybe useful, maybe not 2 Somewhat not useful 1 Extremely not useful

Procedures. Focus groups. Data collection for the local wheelchair service providers will occur in focus groups (4-8 participants per group), either in-person or by Zoom.

On-line survey. The data from global wheelchair service providers will be collected by an online survey that will be self-administered.

End-user interviews. Data collection for the end users will occur individually (wheelchair users with caregivers for Group 1, or wheelchair users alone for Groups 2 and 3), either in-person or remotely.

Data management. The Research Coordinator will use a separate-password-protected tablet or computer to enter all categorical and quantitative data from the focus groups and end-users into a customized REDCap application. Except for the online survey, the interviews will be audio-recorded and transcribed on a laptop computer into Word files using non-cloud-based AI for transcription. Periodic data-validity monitoring will take place. The online questionnaire for wheelchair service providers will also be made available within a REDCap application.

Data analysis. Categorical and quantitative data from each of the three questionnaires will be reported descriptively. The analysis of the qualitative data will be primarily by two investigators, using descriptive coding methodology (that includes the nine steps of data familiarization, developing initial codes, coding the data, refining and revising the codes, categorizing the codes, counting the code frequencies, comparing frequencies across groups, summarizing, and analyzing and reporting findings).

ELIGIBILITY:
Inclusion Criteria:

All participants:

* at least 18 years of age
* willing to participate
* alert
* co-operative
* able to see and hear the video demonstrations
* able to communicate in English
* have the capacity to provide informed consent
* committed to setting a scheduled time for the study activity

Wheelchair service providers:

* Occupational Therapists or Occupational Therapy Assistants who self-identify as being regularly involved in the wheelchair provision process wheelchair users:
* person who has used a manual wheelchair for at least one month caregiving participant:
* spends an average total of at least 2 hours per week with the manual wheelchair user that includes manual wheelchair mobility online survey:
* self-identifies as being regularly involved in the wheelchair provision process

Exclusion Criteria:

• emotional problems that might make participation unsafe or unpleasant

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Local wheelchair service providers will be Occupational Therapists or Occupational Therapy Assistants. Global wheelchair service providers will be people who self-identify as wheelchair service providers. End-users will be wheelchair users and, for some, their caregivers.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-04-15 (Estimated); Primary Completion 2026-04-14 (Estimated); Study Completion 2026-04-14 (Estimated)

PRIMARY OUTCOMES:
Qualitative comments | By 12 months
  For each of a set of problems that have been identified for conventional rear anti-tip devices and a set of potential uses for a new design, study participants will be asked for their subjective comments.

SECONDARY OUTCOMES:
Questions with categorical responses | By 12 months
  For each of a set of problems that have been identified for conventional rear anti-tip devices , study participants will be asked questions for which there are Yes/No answers possible.
Questions with ordinal-scale answers | By 12 months
  For each of a set of potential uses for a new design, study participants will be asked to provide a score from 1-5 on an ordinal scale of potential usefulness.

CONTACTS AND LOCATIONS:
Locations (1):
- Nova Scotia Rehabilitation and Arthritis Centre, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: Yes
Anonymized data will be shared upon request, with the permission of our Research Ethics Board.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: This information will be shared upon request following the approval of the Research Ethics Board, beginning April 15, 2025 and continuing until April 14, 2033.
Access Criteria: University-based researchers will be able to access IPD and supporting material upon request and with the approval of our Research Ethics Board.
URL: https://medicine.dal.ca/departments/department-sites/medicine/divisions/pmr/our-people/faculty/lee-kirby.html